CLINICAL TRIAL: NCT06010784
Title: FUEL: Food, fUn, frEsh, famiLy Program. Improving Children's Diet Through Afterschool Program and Family Support.
Brief Title: 'Food, Fun, Fresh, Family' Program for Healthy Eating and Growth for Elementary-age Children.
Acronym: FUEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Boys & Girls Clubs of the Austin Area (Unknown)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00004545
Record Dates: First submitted 2023-08-18; First posted 2023-08-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Diet, Healthy Growth
Keywords: elementary; after-school program; fruits and vegetable prescription; incentive; produce; school-aged children; family support; CATCH; diet; produce prescription; produce rx; Healthy Eating Index; nutrition incentive; SNAP

STUDY DESIGN:
Intervention Model Description: Community-based trial, two arms randomized on a 1:1 ratio, stratified by SNAP beneficiary status.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research staff responsible for data collection are blinded to the arm allocation of the participant. At the end-point, however, a set of questions about the participant's experience in the program may unblind staff collecting the data. To minimize influence of unblinding, those set of questions will be ask at the end of the data collection period and ensure structured interview techniques are followed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: After-school program + family support (Experimental)
  Interventions: Behavioral: Family support; Behavioral: BGCAA's after-school program with CATCH curriculum
- Control: After-school program only (Active Comparator)
  Interventions: Behavioral: BGCAA's after-school program with CATCH curriculum

INTERVENTIONS:
Behavioral: Family support — * Family tip sheets sent via mobile text at the start of the program and then every 3 weeks, to a total of 6 mobile text messages
  * Weeks 1-4 (4 weeks):
    i. Welcome package mailed in the first week of the program ii. Weekly: one 10-lbs box of produce iii. Recipes accompanying each box (sample recipe card attached to submission) iv. Bi-Weekly: Grocery store gift cards (2x USD 20, to a total of USD 40)
  * Weeks 5-19 (total of 10 weeks over the 19-week study timeline):
    i. An optional online form ("goal sheet") is sent to the parent/caregiver every other week (total 5) with questions about trying new FV items to be submitted in the next 7 days. As an incentive, a USD 10 gift card is sent to those who complete it (a potential total of USD 50).
  ii. Week 11: an extra USD 20 gift card in the week after a school holiday to re-engage participants due to the school-year break.
  Arms: Intervention: After-school program + family support
Behavioral: BGCAA's after-school program with CATCH curriculum — 1. The whole BGCAA's after-school program runs for 3h, Mon-Fri for the school year across all sites where the organization offers the program. All children enrolled are expected to attend a minimum of 2x/week.
  2. In the BGCAA's after-school program, children participate in active recreational time (approx. 60 min, offered 1x/week at a minimum) which is a mixture of free play, structured physical activity games, and/or sports activities (including soccer, football, and basketball).
  3. Uniquely to sites participating in the study, BGCAA's staff will deliver selected CATCH (Coordinated Approach to Child Health) curriculum components in blocks of 45-60 min, 2x/week, as part of the after-school program. The curriculum will focus on healthy eating education and physical activity designed for elementary school-aged children. More information on CATCH at https://catch.org/ (accessed 8/11/2023)

SUMMARY:
The goal of this community-based randomized trial in elementary-aged children and a caregiver (parent/guardian) is to test the effect of providing families with produce and grocery store gift cards (family support) in conjunction with an after-school program for physical activity and healthy eating on improving children's overall diet, in comparison to the child only attending the after-school program without the family support.

Participating families will:

* receive weekly produce bags delivered to their home, recipes, and gift cards to a local grocery store (family support)
* the child will attend the after-school program during the school year

Researchers will compare the child's diet and eating scores with those in the after-school program alone.

DETAILED DESCRIPTION:
Children in grades 1 to 5 and enrolled in after-school program offered by the Boys & Girls Clubs of Austin Area (BGCAA) in selected schools, together with their caregiver (a parent/guardian), will be randomized into one of the two arms:

* Intervention group will receive, for 4 wks, 10 lbs of produce delivered weekly at home and one USD 20 gift card sent bi-weekly (total USD 40). Then, for 15 wks, the caregiver will receive every other week an electronic interactive health goals reminder survey to complete, for which they receive USD10 if completed. The goal sheets are optional activities.
* Control group will receive $120 as grocery store e-gift cards at the end of the study.

Regardless of the allocation arm, the child will attend the BGCAA's afterschool program as part of their family's association with the organization. The program runs daily, and the children are encouraged to attend at least 2x/wk. The "Coordinated Approach to Child Health" (CATCH) program will be delivered as part of the BGCAA program 2x/week.

Primary question: Does a 19-week after-school evidence-based program on nutrition education and physical activity for elementary-aged children improve overall child diet better when resources to encourage healthy eating are also provided to caregivers than when such resources are not provided?

ELIGIBILITY:
Inclusion Criteria:

* Index guardian must be at least 18 years old
* Child must be enrolled in grade 1 to 5 (aged approx. 6-11 y-o) for the 2023-2024 school year
* Child must be enrolled in the BGCAA after-school program at the beginning of the 2023-24 fall semester at one of the 11 sites where BGCAA offers after-school program to elementary school-aged children
* Index parent must be able to speak English and/or Spanish

Exclusion Criteria:

* Already having a sibling enrolled in the study
* Child having serious food allergies or dietary restrictions associated with produce products

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Child's fruit and vegetable intake as measured by the Texas School Physical Activity and Nutrition (TX SPAN) 2019-2020 dietary assessment questions | Baseline, mid-point (4 weeks), end-point (19 weeks)
  This study will use the section of the TX SPAN data collection instrument related to food choices via structured interview (English or Spanish). 32 questions reference specific marker foods or food groups asking the number of times each food group was consumed on the previous day (analogous to a 24h recall), with responses 0 times, 1 time, 2 times or 3 or more times. Total FV variety will be measured by summing the items that ask about fruit and vegetable varieties (excluding juice).
  More on the TX SPAN can be found at <go.uth.edu/SPAN>.
Child's overall diet quality as assessed by SPAN Healthy Eating Index (SHEI) | Baseline, mid-point (4 weeks), end-point (19 weeks)
  As described in 2015 Ranjit et al. SPAN Healthy Eating Index (SHEI) is a composite measure comprising both healthy and unhealthy items from diet measures available in the TX SPAN.
  Healthy score is the sum of previous day consumption of baked or grilled (not fried) meats, milk, yogurt, brown rice, brown pasta, a variety of vegetable types, fruits (not fruit juice), and beans.
  Unhealthy score is the sum of consumption of fried meat, red meat, sugar-sweetened beverages, salty fried snacks, and a variety of dessert items. These are reverse coded, so that the lowest frequency represented the healthiest eating practice.
  These two sums are combined into the single composite SHEI and rescaled from 0-100, where higher scores mean healthier eating practices.

SECONDARY OUTCOMES:
Guardian's fruits and vegetables intake as measured by the NHANES 2009-2010 Dietary Screening Questionnaire (DSQ) | Baseline, mid-point (4 weeks), end-point (19 weeks)
  The DSQ FV module has 10 items that capture frequency of consumption of fruits and vegetables and their sources (such as vegetables in recipes) in the past 30 days. It does not require participants to report serving size. Responses are converted to daily cup equivalent estimates.
BMI-for-age percentile | Baseline, end-point (19 weeks)
  Twice during the program, all children in the after-school program will participate in an interactive activity during a field day where BGCAA staff (blinded to the study arm allocation) measures the children's weight, height and how high they can jump. Because body weight may be a sensitive issue to some children and/or their families, it was proposed to embed it in the daily after-school activities, minimizing the focus on direct and open measurement of weight.
  First, height will be measured using a stadiometer against the wall before the activity. Then, the child will stand on a mat with an integrated scale that will measure their weight. Finally, the children will write their name on an athletic tape and/or post-it notes and jump to stick it to a wall.

OTHER OUTCOMES:
Guardian's mental health as assessed by the Mental Component Score (MCS-12) of the Short-Form 12 Health Survey version 1 (SF-12v1) | Baseline, end-point (19 weeks)
  Self-reported measure assessing the impact of health on an individual's everyday life, often used as a quality of life measure. Two summary scores are reported: 1) a mental component score (MCS-12) and 2) a physical component score (PCS-12). The United States population average PCS-12 is 50 points with standard deviation of 10 points.
Child's mental health status as measured by the Strengths & Difficulties Questionnaire (SDQ) | Baseline, mid-point (4 weeks), end-point (19 weeks)
  SDQ is a brief psychological assessment and behavioral screening tool for 2-17 year-olds (Goodman, 1997), reported by their parents/guardians in the study. 25 items are divided between 5 scales: 1) emotional symptoms (5 items); 2) conduct problems (5 items); 3) hyperactivity/inattention (5 items); 4) peer relationship problems (5 items); 5) prosocial behavior (5 items), with the timeframe of past 6 months. Scores in the sections 1 to 4 are added to generate a total difficulties score (20 items). Higher scores indicate greater difficulties (poorer mental health status).
Child's physical activity engagement as measured by the physical activity questions in the Texas School Physical Activity and Nutrition (TX SPAN) 2nd grade 2019-2020 | Baseline, end-point (19 weeks)
  Questions are posed to the guardian. Two items assess 1) how many days in the past week the child was physically active for at least 60 min. and 2) played outdoors for at least 30 min. outside of school hours. The other 5 items assess attitude and usual engagement in physical activity. The demographics survey at baseline will ask whether the child has limited physical ability to engage in activities.

CONTACTS AND LOCATIONS:
Overall Officials: Maninder Kahlon, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Boys & Girls Clubs of Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
By request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT06010784/Prot_SAP_001.pdf